CLINICAL TRIAL: NCT03587636
Title: Prospective Randomized Controlled Trial Comparing Liposomal Bupivacaine to Bupivacaine Interscalene Blocks for Total Shoulder Arthroplasty Surgery; a Pilot Study
Brief Title: Liposome Bupivacaine Interscalene Total Shoulder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ANES-2018-26661
Record Dates: First submitted 2018-06-20; First posted 2018-07-16 (Actual); Results first posted 2022-05-02 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Acute Pain
MeSH Terms: conditions — Acute Pain | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Liposome bupivacaine interscalene block (Experimental): 10 mL of liposome bupivacaine and 10 mL of 0.5% bupivacaine will be injected at the interscalene brachial plexus under ultrasound guidance
  Interventions: Drug: liposome bupivacaine
- bupivacaine interscalene block (Active Comparator): 20 mL of 0.5% bupivacaine will be injected at the interscalene brachial plexus under ultrasound guidance.
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: liposome bupivacaine — interscalene block with liposomal bupivacaine plus bupivacaine
  Other Names: bupivacaine
  Arms: Liposome bupivacaine interscalene block
Drug: Bupivacaine — interscalene block with bupivacaine
  Arms: bupivacaine interscalene block

SUMMARY:
This is a randomized prospective outcomes study comparing two groups of patients. One group will receive liposomal bupivacaine plus bupivacaine and the other will receive bupivacaine alone in interscalene blocks when undergoing total shoulder arthroplasty. The purpose of the study is to determine if LB plus bupivacaine provides superior pain control compared to bupivacaine alone when injected in an interscalene block for patients undergoing total shoulder arthroplasty surgery.

DETAILED DESCRIPTION:
Liposomal bupivacaine (LB) is a long acting local anesthetic. It is liposome encapsulated bupivacaine which allows for prolonged release of bupivacaine over a 72-hour period. Bupivacaine is a medium acting local anesthetic which provides between 6 and 24 hours of analgesia when used in a peripheral nerve block. Both medications are standard of care for use in interscalene blocks here at the U of MN.

LB has not been adequately studied in peripheral nerve blocks and has yet to be studied for use in interscalene blocks for Total Shoulder Arthroplasty (TSA) patients. It has been studied in Rotator Cuff Repairs (RCR) surgery and showed superior analgesia compared to bupivacaine.

The purpose of the study is to determine if LB plus bupivacaine provides superior pain control compared to bupivacaine alone when injected in an interscalene block for patients undergoing total shoulder arthroplasty surgery.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients aged greater than 18 years of age that are undergoing total or reverse total shoulder arthroplasty

Exclusion Criteria:

* Patients with allergy to local anesthetics, daily use of opioids for more than 3 weeks prior to surgery, patient refusal, patient with coagulopathy, non-english speaking patients, and those who do not have access to a telephone.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2018-09-17 (Actual); Primary Completion 2021-03-15 (Actual); Study Completion 2021-03-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Flaherty, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment ceased after 70 patients completed the study per protocol
Period: Overall Study
Arm/Group | Bupivacaine Interscalene Block | Liposome Bupivacaine Interscalene Block
Started | 39 | 38
Completed | 37 | 33
Not Completed | 2 | 5
Not completed — Lost to Follow-up | 2 | 5

BASELINE CHARACTERISTICS:
Population: Total of 75 included here due to dropouts along the way
Groups:
- Total: Total of all reporting groups
Arm/Group | Bupivacaine Interscalene Block | Liposome Bupivacaine Interscalene Block | Total
Number analyzed (Participants) | 38 | 37 | 75
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 14 | 29
  >=65 years | 23 | 23 | 46
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 15 | 37
  Male | 16 | 22 | 38
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Total Opioid Use
Description: total amount of opioid use from after surgery through 72 hours. Opioids normalized to morphine equivalents
Time Frame: From end of surgery through 72 hours after end of surgery
Measure: Median (Inter-Quartile Range); unit: mg (morphine equivalent)
Arm/Group | Bupivacaine Interscalene Block | Liposome Bupivacaine Interscalene Block
Number analyzed (Participants) | 37 | 33
mg (morphine equivalent) | 22.5 [7.5 to 96.0] | 30.0 [5.6 to 45.0]

2. Secondary Outcome: Total Maximum Pain Scores f
Description: Sum total of maximal pain scores through 72 horus after surgery. Pain scores reported on a numerical rating scale from 0-10. 10 is worse and 0 is best
Time Frame: time from end of surgery through 72 hours after end of surgery
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Bupivacaine Interscalene Block | Liposome Bupivacaine Interscalene Block
Number analyzed (Participants) | 37 | 33
score on a scale | 4.0 [2.0 to 6.0] | 3.0 [1.0 to 5.5]

ADVERSE EVENTS:
Time Frame: 72 hours
Arm/Group | Bupivacaine Interscalene Block | Liposome Bupivacaine Interscalene Block
All-Cause Mortality (participants affected / at risk) | 0/37 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/33
Other Adverse Events (participants affected / at risk) | 7/37 | 0/33
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bupivacaine Interscalene Block (N=37) | Liposome Bupivacaine Interscalene Block (N=33)
Fall weeks after surgery (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Balance Issues weeks after surgery (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Numbness/ swelling (Nervous system disorders) | 1 (1) | 0 (0)
Bruising/ swelling (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Appendicitis several weeks after surgery (Infections and infestations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-06-03): https://cdn.clinicaltrials.gov/large-docs/36/NCT03587636/Prot_SAP_000.pdf
  • Informed Consent Form (2020-03-26): https://cdn.clinicaltrials.gov/large-docs/36/NCT03587636/ICF_001.pdf